CLINICAL TRIAL: NCT05317975
Title: The Cardiopulmonary Function Outcome and the Effect of Two Modules of Home-based Rehabilitation Programs in Patients After COVID-19 Infection - A Randomized and Controlled Trial.
Brief Title: The Effect of Home-based Rehabilitation Program After COVID-19 Infection
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Recruitment difficulties and insufficient funding.
Sponsor: National Taiwan University Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 202106093RIND
Record Dates: First submitted 2022-03-31; First posted 2022-04-08 (Actual); Last update posted 2025-02-19 (Actual); Status verified 2025-02

CONDITIONS: COVID-19
Keywords: COVID-19; Rehabilitation; Cardiopulmonary exercise testing
MeSH Terms: conditions — COVID-19

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Add-on telerehabilitation combined with usual home-based rehabilitation (Experimental): Add-on telerehabilitation combined with usual home-based rehabilitation
  Interventions: Behavioral: Add-on telerehabilitation and home-based rehabilitation
- Stand-alone usual home-based rehabilitation (Experimental): Stand-alone usual home-based rehabilitation
  Interventions: Behavioral: Home-based rehabilitation alone
- Usual care (No Intervention): Usual care

INTERVENTIONS:
Behavioral: Add-on telerehabilitation and home-based rehabilitation — 1. 12wk home-based rehabilitation including individualized exercise training and inspiratory muscle training with symptoms monitoring. Participants will be provided with a manual and routine telephone follow-up by a case manager.
  2. Add-on telerehabilitation for instruction and supervision of exercise training
  Arms: Add-on telerehabilitation combined with usual home-based rehabilitation
Behavioral: Home-based rehabilitation alone — 12wk home-based rehabilitation including individualized exercise training and inspiratory muscle training with symptoms monitoring. Participants will be provided with a manual and routine telephone follow-up by a case manager.
  Arms: Stand-alone usual home-based rehabilitation

SUMMARY:
To follow up the cardiopulmonary function after coronavirus disease 2019 (CoVID-19) infection and compare the effect of a 12-week home-based cardiopulmonary with or without add-on remote rehabilitation on the cardiopulmonary function, emotion and quality of outcome.

DETAILED DESCRIPTION:
The investigators will recruit the patients post-CoVID infection for a cardiopulmonary function evaluation and a home-based rehabilitation program. The investigators hypothesize that an add-on remote rehabilitation on a home-based rehabilitation has a better effect than a home-based rehabilitation alone on the compliance rate for the exercise, and also a better outcome in terms of cardiopulmonary function testing, 6-minute walking test, physical activities and quality of life, as well as less dyspnea, depression and anxiety.

ELIGIBILITY:
Inclusion criteria:

1. ≥ 20 years of age.
2. COVID-19 survivor after de-isolation at post-acute stage about to be discharged or already at outpatient follow-up who still have symptoms or exercise intolerance.

Exclusion criteria:

1. Unable to cooperate with rehabilitation or evaluation.
2. Dependent in basic activities of living before infection (Premorbid Barthel index <80).
3. End stage patient, with life expectancy less than 1 year.
4. Having contraindications for exercise according to the evaluation of a physician.

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 13 (Actual)
Dates: Start 2021-07-15 (Actual); Primary Completion 2024-02-17 (Actual); Study Completion 2025-02-17 (Actual)

PRIMARY OUTCOMES:
Change of 6-minute walking test (6MWT) and exercise capacity | The change in 6MWT and peak oxygen uptake will be measured at baseline, 12 weeks, 6 and 12 months after intervention.
  The distance of a 6-minute walking test and peak oxygen uptake according to cardiopulmonary exercise test will be assessed before intervention (12-week rehabilitation course), 12 weeks, 6 months and 12 months after intervention.

SECONDARY OUTCOMES:
Dyspnea scale | The change in mMRC will be measured at baseline, 12 weeks, 6 and 12 months after intervention.
  The investigators will assess the change in the Modified Medical Research Council (mMRC) scale. The mMRC scale ranges from 0 to 4. Higher scores indicate worsen symptoms.
Fatigue | The change in BFI will be measured at baseline, 12 weeks, 6 and 12 months after intervention.
  The investigators will assess the change in the Brief Fatigue Inventory (BFI). The total score of BFI ranges from 0 to 10. Higher scores indicate greater level of fatigue.
Depression and anxiety | The change in PHQ-9 and GAD-7 will be measured at baseline, 12 weeks, 6 and 12 months after intervention.
  The investigators will assess the change in Patient Health Questionnaire (PHQ-9) and Generalized Anxiety Disorder scale (GAD-7). The PHQ-9 score ranges from 0-27 and the GAD-7 score ranges 0-21. Higher scores indicate worsen symptoms.
Cognitive evaluation | The change in MoCA will be measured at baseline, 12 weeks, 6 and 12 months after intervention.
  The investigators will assess the change in Montreal Cognitive Assessment (MoCA). The total score of MoCA ranges from 0 to 30. Higher scores indicate better cognitive function.
Quality of life evaluation | The change in EQ-5D will be measured at baseline, 12 weeks, 6 and 12 months after intervention.
  The investigators will assess the change in EuroQol-5D.
Grip strength | The change in grip strength will be measured at baseline, 12 weeks, 6 and 12 months after intervention.
  The investigators will assess the grip strength using a grip goniometer with the participants seated and the elbow flexed at 90 degree.

CONTACTS AND LOCATIONS:
Overall Officials: Hung-Jui Chuang, MD, Principal Investigator — Department of Physical Medicine and Rehabilitation, National Taiwan University Hospital
Locations (1):
- National Taiwan University Hospital, Taipei, Taiwan

IPD SHARING:
Plan to Share IPD: No